CLINICAL TRIAL: NCT02744378
Title: Comparison of Tacrolimus 0.1% and Clobetasol 0.05% in the Management of Symptomatic Oral Lichen Planus- A Double-blinded Randomized Clinical Trial in Sri Lanka
Brief Title: Comparison of Tacrolimus 0.1% and Clobetasol 0.05% in the Management of Symptomatic Oral Lichen Planus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Peradeniya (Other)
Responsible Party: Principal Investigator, Dr. P.V.K.S Hettiarachchi, Dr, University of Peradeniya
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RG/2013/08/D
Record Dates: First submitted 2016-04-06; First posted 2016-04-20 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Oral Lichen Planus
MeSH Terms: conditions — Lichen Planus, Oral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clobetasol Group (Active Comparator): clobetasol propionate (0.05%) cream
  Interventions: Drug: Clobetasol 0.05%
- Tacrolimus Group (Active Comparator): tacrolimus (0.1%) cream
  Interventions: Drug: Tacrolimus 0.1%

INTERVENTIONS:
Drug: Tacrolimus 0.1% — This group was randomly allocated to receive topical Tacrolimus 0.1% for 3 consecutive weeks
  Arms: Tacrolimus Group
Drug: Clobetasol 0.05% — This group was randomly allocated to receive topical Clobetasol 0.05% for 3 consecutive weeks
  Arms: Clobetasol Group

SUMMARY:
This clinical study is carried out to assess the efficacy of Tacrolimus and Clobetasol in symptomatic Oral Lichen Planus.

ELIGIBILITY:
Inclusion Criteria:

* Clinically and Histologically proven Oral Lichen Planus
* Symptomatic

Exclusion Criteria:

* topical/ systemic medication for OLP in the previous three months
* contraindication for medications use such as a history of allergy to either corticosteroids/ tacrolimus
* immunosuppression, or pregnant / lactating females
* lichenoid reactions either drug induced or due to dental amalgam
* diabetes mellitus and on oral hypoglycemic drugs
* systemic involvement such as concurrent skin/genital lesions

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-06; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The intensity of Pain | Three weeks after the application of drugs
  The intensity of pain was assessed using visual analog scale (VAS) - The patients were asked to score their intensity of pain using a VAS where the pain scores ranged from 0 (no pain) to 10 (extreme pain)
  Four VAS was recorded one for spicy food and the other one for without spicy food for right side and left sides separately. The mean VAS was calculated for each side and the severity of pain was evaluated according to the following scales:
  Scale 0: no pain: VAS=0, Scale 1: mild pain: 0< VAS≤3.5, Scale 2: moderate pain: 3.5 <VAS≤7, Scale 3: severe pain: 7< VAS≤10.
The clinical response | Three weeks after the application of drugs
  The clinical response of the lesion was scored according to the grading system formulated by Thongprasom et al.,in 1992 for the mucosal lesions:
  Score 5 = white striae with erosive area more than 1 cm, Score 4 = white striae with erosive area less than 1 cm, Score 3 = white striae with atrophic area more than 1 cm, Score 2 = white striae with atrophic area less than 1 cm, Score 1 =mild white striae, no erythematous area Score 0 = no lesion, normal mucosa. This scorings were performed for both right and left sides separately.